CLINICAL TRIAL: NCT03856333
Title: Determining the Validity, Reliability and Responsiveness of Cognitive Exercise Therapy Approach Scale in Patients With Chronic Neck Pain
Brief Title: Cognitive Exercise Therapy Approach Scale in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özge Şahin, physiotherapist, Eastern Mediterranean University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OZ 1313
Record Dates: First submitted 2019-02-18; First posted 2019-02-27 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Evaluation; Treatment
Keywords: Cognitive Exercise Therapy Approach Scale; validity; reliability; responsiveness; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- traditional treatment (Other): 30 minutes of conventional TENS, 20 minutes of hotpack, 8 minutes of therapeutic ultrasound and isotonic, isometric, stretching and relaxation exercises 2 weeks, 5 days in a week.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — exercises, physical agents

SUMMARY:
The aim of this study was to determine the validity, reliability and sensitivity of the Cognitive Exercise Therapy Approach Scale in patients with neck pain.

DETAILED DESCRIPTION:
According to the power analyzes 199 neck pain patients will be taken to the study.The study will be initiated after the approval of the Ethics Committee of the Eastern Mediterranean University Faculty of Health Sciences. After informing about the content of the study, individuals who want to participate in the study will be asked to sign the informed consent form. In order to evaluate the validity and reliability of the BETY scale in the study, the same individuals will be given a test-retest with 1 week intervals. In these tests, the Neck Disability Index (NDI), Arm Shoulder and Hand Problems Questionnaire (DASH), Short Form-36 (SF-36), Hospital Anxiety and Depression Scale (HADS) and BETY scale will be applied.In order to assess the sensitivity to change, 44 individuals will be asked to re-fill the forms after the traditional physiotherapy program for neck pain, which will be administered 10 sessions. For 2 weeks, a routine exercise program consisting of 20 minutes of conventional TENS, 20 minutes of hotpack, 8 minutes of therapeutic ultrasound and isotonic, isometric, stretching and relaxation exercises will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-65 years
* Neck pain VAS out of 3 and above which individuals
* Individuals who have neck pain for more than 3 months

Exclusion Criteria:

* Patients with previous neck surgery history
* Not willing to participate in the study
* Attract trouble understanding for filling scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach Scale (BETY) | Change from the baseline will be assesed at the first week and at the third week.
  The biopsychosocial process associated with the neck pain will be evaluated by the 'Cognitive Exercise Therapy Approach Scale'.
  The scale consists of 30 items. The scale was scored using a 5-point Likert system. Every question; No in no time: 0, Yes rarely: 1, Yes sometimes: 2, Yes often: 3, Yes is always scored as 4: and gives a total score of 30 items. High score means low biopsychosocial status assessment is "bad

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | At the beginning and 2 weeks after the start of treatment
  It is used to assess the disability caused by neck pain. The index consists of 10 chapters including the severity of pain, personal care, lifting, reading, headache, concentration, working life, driving, sleep and leisure time. There are 6 responses for each section, 0 (no pain and no functional limitation) and 5 (worst pain and maximum limitation). There was no apology between 0-4 points in the NDI, mild disability between 5-14 points, moderate disability between 15-24 points, severe apology between 25-34 points and full disability over 35 points . The Turkish validity and reliability study was conducted by Aslan et al.
Arm, Shoulder and Hand Problems Questionnaire (DASH) | At the beginning and 2 weeks after the start of treatment
  It is a scale used to evaluate the functional disability associated with upper extremity. The scale consists of three parts. DASH has a total of 30 questions and includes 8 questions for people who are engaged in work and social activities. In case of not answering more than 3 questions, the questionnaire is considered invalid. Response options in scale are between 1 and 5. Scoring for each section is calculated as 0-100. High scores indicate serious activity limitations . The scale is valid, reliable and sensitive to changes. The Turkish cultural adaptation was also made and the scale was found to be valid and reliable for the Turkish version.
Hospital Anxiety and Depression Scale (HADS) | At the beginning and 2 weeks after the start of treatment
  The area of use of the scale is not to diagnose, but to reveal the depression and anxiety associated with existing diseases. It has been widely used in a variety of somatic, psychiatric and primary care populations and in many chronic diseases such as musculoskeletal, cancer, end-stage renal disease, and has been found to be able to measure depression and anxiety significantly . It is a 14-item scale consisting of seven anxiety-related subscales (HADS-A) and depression subscale (HADS-D). Each question is scored between 0 and 3 and is interpreted according to the total score. Although the total score indicates the increased level of anxiety and depression, it can be interpreted as being 'normal' between 0-7, being between 8-10, 'borderline normal', and between 11-21 being 'abnormal'. The Turkish validity and reliability study was conducted by Aydemir et al.
Short Form-36 (SF-36) | At the beginning and 2 weeks after the start of treatment
  This questionnaire, which evaluates the quality of life of the person, consists of 36 questions on eight sub-scales: physical function, physical role restriction, emotional role restriction, body pain, social function, mental health, vitality, and general health. The scores are scored separately for each subscale and the scores range from 0 to 100. 100 points indicate good health status, while 0 points indicate poor health status . The reliability and validity study of Turkish by Koçyiğit et al .
Visual Analogue Scale (VAS) | At the beginning, and 2 weeks after the start of treatment
  The pain intensity of individuals was questioned by Vizel Analog Scale. VAS is a method used in numerical form to quantify non-measured values. It is often preferred because it can be easily applied and repeated in a short time. The parameter to be evaluated in a horizontal line of 10 centimeters is written to define both endpoints and the patient is asked to mark the appropriate point for the parameter evaluated on this 10-centimeter line. The severity of the patient's pain is determined by measuring the length of the distance from the point of pain to the point determined by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Özge Şahin, Principal Investigator — EMU; Sevim Öksüz, PhD, Study Director — EMU; Ender Angın, PhD, Study Director — EMU
Locations (1):
- Özge Şahin, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No
Not ethical